CLINICAL TRIAL: NCT05134493
Title: Embolic Signals Detection Study (Esds) in Candidates for Surgical Carotid Revascularisation: a Comparison With Plaque Histological Findings
Brief Title: Embolic Signals Detection Study (Esds) in Candidates for Surgical Carotid Revascularisation
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, Ginevra Pizzarelli, Dr. Ginevra Pizzarelli, Medico in Formazione Specialistica, Azienda Ospedaliero-Universitaria di Modena
Other Study IDs: 176/2018/OSS/AOUMO - MESTCD
Record Dates: First submitted 2021-06-25; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Carotid Stenosis; Carotid Artery Diseases; Carotid Atherosclerosis; Carotid Artery Plaque; TCD; Stroke
Keywords: carotid; carotid stenosis; plaque; stroke risk; transcranial doppler; TCD; histology
MeSH Terms: conditions — Carotid Stenosis; Carotid Artery Diseases; Stroke; Plaque, Amyloid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — carotid plaque
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
About 20% of strokes are caused by emboli deriving from a carotid plaque. In symptomatic patients with carotid stenosis grater than 70% the Carotid Endarterectomy (CEA) reduces stroke risk by about 75% and is generally accepted as being cost effective. However also in these cases there is a part of the population that, according to the morphological plaque characteristics, could better benefit from a conservative medical treatment.

Improving the Best Medical Treatment, the situation seems to be even less clear in asymptomatic patients, where probably it would need to treat at least 32 patients in order to prevent one single ictus.

Different parameters have been considered in order to determine, among the asymptomatic patients the ones that more than others could benefit from a surgical revascularisation instead of a medical treatment.

Between these parameters, the quality of the plaque (vulnerability) and the micro-embolic signals (MES) detection with the Transcranial Doppler (TCD) Holter seems to be the most relevant.

Another interesting aspect is trying to establish whether plaques can determine a different embolic risk in relation to the different histological findings.

Therefore, it seems interesting and reasonable trying to establish a correlation between these two parameters in asymptomatic patients as in the symptomatic ones in order to make more and more appropriate a surgical plaque removal according to the specific risk of each patient in a set of tailored surgery.

It consists in a descriptive observational study, since it intends to describe the embolic signals detection (MES) counted in automatic way with the TCD Holter, in patients affected by carotid stenosis, before and after the surgical operation.

In particular it consists in a monocentric, longitudinal, prospective cohort study since it intends to analyse a group of patients (already candidates to CEA) that experiences a specific event (MES) before and after the surgical plaque removal, in a precise span of time.

Since the treatment, removing the plaque, should remove the embolic focus too, a significant reduction of microembolic signals in post-operative time is expected.

This reduction has been esteemed around about the 70% among candidates to CEA. Patients taken on responsibility of the equipe will undergo an ultrasonographic investigation for the carotid stenosis, histological characterization of the plaque based on the Gray-Weale classification and TCD-Holter for MES.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed
* Age>18y.o.
* Carotid stenosis >70% and/or vulnerable plaque

Exclusion Criteria:

* Inability to give the informed consent
* Age<18y.o.
* Carotid stenosis < 70 %
* Patients already treated with CEA in the same seat
* Impossibility to find the insonation window
* Patients not in best medical treatment therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We selected patients already got in touch with the hospital, already put in list for a carotid surgical revascularization.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
MES COUNT | before surgery
  number of MES
MES COUNT | 24 hours after surgery
  number of MES
MES COUNT | after 30 days from the surgery
  number of MES

SECONDARY OUTCOMES:
RISK RATE | through study completion, an average of 60 days
  Estimate an association between MES count and plaque's histology

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Moratto, Dr, Principal Investigator — AOU Modena e Reggio Emilia
Locations (1):
- OCB Baggiovara, AOU Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pizzarelli G, Gennai S, Leone N, Covic T, Moratto R, Silingardi R. Transcranial Doppler detects micro emboli in patients with asymptomatic carotid stenoses undergoing endarterectomy. J Vasc Surg. 2023 Mar;77(3):811-817.e2. doi: 10.1016/j.jvs.2022.10.003. Epub 2022 Oct 13. PMID 36243263